CLINICAL TRIAL: NCT07175948
Title: Outcome of Different Clinical Phenotypes of Myocarditis in Children Admitted to Assiut University Children Hospital
Brief Title: Outcome of Clinical Phenotypes of Pediatric Myocarditis at Assiut University Children Hospital
Acronym: PED-MYO
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elshymaa Abdelmged Abdelmenaem, resident , pediatric department, Assiut University
Other Study IDs: AUMCH-MYO-2025
Record Dates: First submitted 2025-09-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Myocarditis; Myocarditis Acute
Keywords: Viral Myocarditis; Cardiogenic Shock
MeSH Terms: conditions — Myocarditis; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute Myocarditis: Children (1-18 years) diagnosed with acute myocarditis, typically following viral illness, presenting with fever, chest pain, heart failure symptoms, or arrhythmias. Diagnosis supported by elevated cardiac biomarkers, echocardiographic findings of LV dysfunction, and ECG changes. Management includes standard medical therapy (inotropes, ACE inhibitors, beta-blockers) and in some cases corticosteroids or IVIG depending on severity.
  Interventions: Other: Standard Medical Therapy; Drug: Standard Medical Therapy
- Fulminant Myocarditis: Children presenting with sudden, severe myocarditis characterized by rapid onset of cardiogenic shock, severe LV dysfunction, or multi-organ involvement. Diagnosis based on clinical picture, elevated biomarkers, echocardiography, and ECG. Management frequently requires intensive care, high-dose inotropes, and may include IVIG, corticosteroids, and mechanical circulatory support such as ECMO if indicated.
  Interventions: Other: Standard Medical Therapy; Drug: Standard Medical Therapy
- Chronic Active Myocarditis: Children with ongoing inflammatory myocarditis lasting weeks to months, presenting with persistent heart failure symptoms, arrhythmias, or progressive LV dysfunction. Diagnosis confirmed by echo and biomarkers, sometimes MRI. Treatment includes standard therapy for heart failure plus immunomodulation with corticosteroids and/or IVIG in selected cases. Close monitoring is required to prevent progression.
  Interventions: Other: Standard Medical Therapy; Drug: Standard Medical Therapy
- Chronic Persistent Myocarditis: Children with a long-term, indolent course of myocarditis, often progressing toward dilated cardiomyopathy. Patients present with signs of chronic heart failure, reduced EF, and persistent LV dilation. Management includes conventional heart failure therapy (ACE inhibitors, beta-blockers, diuretics, inotropes as needed). Corticosteroids or IVIG may be used in selected patients based on clinical status. Long-term follow-up is required.
  Interventions: Other: Standard Medical Therapy; Drug: Standard Medical Therapy

INTERVENTIONS:
Other: Standard Medical Therapy — All enrolled children will receive standard medical therapy tailored to clinical status. This includes inotropes (e.g., dopamine, dobutamine, milrinone), ACE inhibitors, beta-blockers, and/or diuretics as indicated. Treatment is supportive and adjusted according to severity of cardiac dysfunction and hemodynamic status. The goal is to stabilize heart failure, improve cardiac output, and prevent progression to dilated cardiomyopathy.
Drug: Standard Medical Therapy — All enrolled children will receive standard medical therapy tailored to clinical status. This includes inotropes (dopamine, dobutamine, milrinone), ACE inhibitors, beta-blockers, and/or diuretics as indicated. Therapy is supportive and adjusted according to severity of cardiac dysfunction and hemodynamic status to stabilize heart failure, improve cardiac output, and prevent progression to dilated cardiomyopathy.
  2️⃣ Intervention 2

SUMMARY:
This study aims to investigate the clinical phenotypes, management approaches, and outcomes of myocarditis in children admitted to Assiut University Children's Hospital. Myocarditis is an inflammatory disease of the heart muscle that can present in different clinical forms, including acute, fulminant, chronic active, and chronic persistent types. These forms vary in severity, treatment needs, and long-term outcomes.

Children aged 1-18 years who are diagnosed with myocarditis based on clinical findings, cardiac biomarkers, echocardiography, and electrocardiography (with MRI when available) will be included. Patients with congenital heart disease or cardiomyopathy unrelated to myocarditis will be excluded.

The study will follow eligible patients prospectively over a 12-month period. Detailed clinical assessment, laboratory tests, echocardiographic findings, and management strategies will be recorded. Special attention will be given to the role of corticosteroids and intravenous immunoglobulin (IVIG) in treatment. Outcomes including recovery of cardiac function, need for intensive care, and survival will be assessed.

By analyzing the clinical presentation, treatment, and prognosis of different myocarditis phenotypes, this study aims to improve the understanding of disease patterns in children and provide evidence to guide future management.

DETAILED DESCRIPTION:
Myocarditis is an inflammatory disorder of the myocardium that may cause myocyte injury, necrosis, and cardiac dysfunction. Pediatric myocarditis has heterogeneous clinical phenotypes, commonly categorized into acute, fulminant, chronic active, and chronic persistent forms. These categories differ in pathophysiology, clinical presentation, and prognosis, making phenotypic classification essential for guiding treatment decisions and predicting outcomes.

In children, acute myocarditis often follows viral infection and may manifest with fever, chest pain, palpitations, or signs of heart failure. Fulminant myocarditis presents abruptly with severe hemodynamic compromise and cardiogenic shock, requiring intensive care and often mechanical circulatory support. Chronic active myocarditis is associated with ongoing inflammation, progressive ventricular dysfunction, and increased risk of dilated cardiomyopathy. Chronic persistent myocarditis may present with milder, prolonged symptoms but can still result in long-term morbidity.

This prospective cohort study will be conducted at Assiut University Children's Hospital over 12 months. Approximately 30 eligible pediatric patients will be enrolled using consecutive sampling. Inclusion criteria include children aged 1-18 years with clinically and diagnostically confirmed myocarditis. Exclusion criteria include congenital heart disease or cardiomyopathy unrelated to myocarditis.

All participants will undergo comprehensive evaluation including:

Clinical assessment: demographic data, presenting symptoms, signs of cardiac dysfunction, and general/systemic examination.

Laboratory tests: cardiac biomarkers (troponin, CK-MB), inflammatory markers (CRP, ESR), renal and liver function, lactate, and ABG.

Echocardiography: left ventricular dimensions, fractional shortening, ejection fraction, wall motion abnormalities, pericardial effusion, and valve regurgitation.

Electrocardiography and chest X-ray.

Management recording: medical therapy including corticosteroids, IVIG, inotropes, and supportive care.

Primary outcomes: classification of myocarditis phenotypes and assessment of treatment effectiveness, with focus on corticosteroids and IVIG.

Secondary outcomes: clinical improvement, recovery of cardiac function, survival, and requirement of intensive care or mechanical circulatory support.

Statistical analysis will be performed using SPSS. Data will be analyzed using descriptive and analytical methods, including Chi-square, t-tests, correlation, and regression analyses, with significance set at p < 0.05.

This study will contribute to understanding the spectrum of pediatric myocarditis in a tertiary care setting in Upper Egypt and provide insight into prognostic indicators and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* • Children aged between 1 to 18 years.

  * Children diagnosed with myocarditis based on clinical presentation, echocardiography, and cardiac biomarkers, ECG and MRI (if available)

Exclusion Criteria:

* • Children with congenital heart disease.

  * Known cardiomyopathy unrelated to myocarditis.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All available patients diagnosed with myocarditis and attending Assiut University children hospital during the study period will be included in this study All patients included in the study will have fulfilled the established criteria to ensure the appropriateness and consistency of the study population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Classification of clinical phenotypes of myocarditis in children | At baseline (study enrollment, within first hospital visit).
  Phenotypic classification (acute, fulminant, chronic active, chronic persistent) will be assigned based on clinical presentation, echocardiography, cardiac biomarkers, and ECG/MRI findings.
Classification of clinical phenotypes of myocarditis in children | At baseline (upon parental enrollment, assessed once at study start).
  Phenotypic classification (acute, fulminant, chronic active, chronic persistent) will be assigned based on clinical presentation, echocardiography, cardiac biomarkers, and ECG/MRI findings.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao Q, Zhan S. Corticosteroid in anti-inflammatory treatment of pediatric acute myocarditis: a systematic review and meta-analysis. Ital J Pediatr. 2023 Mar 13;49(1):30. doi: 10.1186/s13052-023-01423-w. PMID 36915162
- [Background] Hajjar LA, Teboul JL. Mechanical Circulatory Support Devices for Cardiogenic Shock: State of the Art. Crit Care. 2019 Mar 9;23(1):76. doi: 10.1186/s13054-019-2368-y. PMID 30850001
- [Background] Kociol RD, Cooper LT, Fang JC, Moslehi JJ, Pang PS, Sabe MA, Shah RV, Sims DB, Thiene G, Vardeny O; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology. Recognition and Initial Management of Fulminant Myocarditis: A Scientific Statement From the American Heart Association. Circulation. 2020 Feb 11;141(6):e69-e92. doi: 10.1161/CIR.0000000000000745. Epub 2020 Jan 6. PMID 31902242
- [Background] Jayashree M, Patil M, Benakatti G, Rohit MK, Singhi S, Bansal A, Baranwal A, Nallasamy K, Angurana SK. Clinical Profile and Predictors of Outcome in Children with Acute Fulminant Myocarditis Receiving Intensive Care: A Single Center Experience. J Pediatr Intensive Care. 2021 Jan 25;11(3):215-220. doi: 10.1055/s-0040-1722339. eCollection 2022 Sep. PMID 35928042
- [Background] Garbern JC, Gauvreau K, Blume ED, Singh TP. Is Myocarditis an Independent Risk Factor for Post-Transplant Mortality in Pediatric Heart Transplant Recipients? Circ Heart Fail. 2016 Jan;9(1):e002328. doi: 10.1161/CIRCHEARTFAILURE.115.002328. Epub 2015 Dec 23. PMID 26699389
- [Background] Ammirati E, Frigerio M, Adler ED, Basso C, Birnie DH, Brambatti M, Friedrich MG, Klingel K, Lehtonen J, Moslehi JJ, Pedrotti P, Rimoldi OE, Schultheiss HP, Tschope C, Cooper LT Jr, Camici PG. Management of Acute Myocarditis and Chronic Inflammatory Cardiomyopathy: An Expert Consensus Document. Circ Heart Fail. 2020 Nov;13(11):e007405. doi: 10.1161/CIRCHEARTFAILURE.120.007405. Epub 2020 Nov 12. PMID 33176455
- [Background] Lasica R, Djukanovic L, Savic L, Krljanac G, Zdravkovic M, Ristic M, Lasica A, Asanin M, Ristic A. Update on Myocarditis: From Etiology and Clinical Picture to Modern Diagnostics and Methods of Treatment. Diagnostics (Basel). 2023 Sep 28;13(19):3073. doi: 10.3390/diagnostics13193073. PMID 37835816
- [Background] P. Shakuntala and V. Sumitra, "Acute Myocarditis," Indian Journal of Practical Pediatrics, vol. 10, no. 2, pp. 65-73, Apr. 2025,
- See also: Official website of Assiut University Faculty of Medicine, host institution for this study. — https://www.aun.edu.eg/medicine